CLINICAL TRIAL: NCT06466031
Title: Application of MET-PET in Fusion With MRI in the Surgical Treatment and Postoperative Radiotherapy of Glioblastoma Multiforme - a Randomized, Blinded, Prospective Study
Brief Title: Application of MET-PET in Fusion With MRI in the Treatment of Glioblastoma Multiforme
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Copernicus Memorial Hospital (Other)
Collaborators: Medical Research Agency, Poland (Other Government)
Responsible Party: Principal Investigator, Kamil Krystkiewicz, Principal Investigator, Copernicus Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023/ABM/01/00010
Record Dates: First submitted 2024-06-02; First posted 2024-06-20 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Glioblastoma Multiforme
Keywords: Glioblastoma Multiforme; Methionine; Positron-Emission Tomography; Brain neoplasms; Progression-free survival; Dose Fractionation, Radiation; Post-surgical radiotherapy
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Resection and radiotherapy according to the MRI & PET fusion (Experimental): Tumor resection and radiotherapy will be planned based on the fusion of MRI and PET.
  Interventions: Other: MRI & PET fusion
- Radiotherapy according to the MRI & PET fusion (Experimental): Tumor resection will be planned based on the MRI. Radiotherapy will be planned according to the fusion of MRI & PET.
  Interventions: Other: MRI & PET fusion; Other: MRI+T1C
- Resection and radiotherapy according to the MRI (Sham Comparator): Tumor resection and radiotherapy will be planned based on the MRI.
  Interventions: Other: MRI+T1C

INTERVENTIONS:
Other: MRI & PET fusion — MRI+T1C in fusion with MET-PET will be used for tumor resection and/or radiotherapy planning. Resection will be terminated after removal of PET-assigned tumor margin or in case any neuromonitoring-based indications regarding neurological damage occur.
  Arms: Radiotherapy according to the MRI & PET fusion; Resection and radiotherapy according to the MRI & PET fusion
Other: MRI+T1C — MRI+T1C will be used for tumor resection and radiotherapy planning. Resection will be terminated after removal of contrast-enhancing part regardless of 5-ALA fluorescence or in case any neuromonitoring-based indications regarding neurological damage occur.
  Arms: Radiotherapy according to the MRI & PET fusion; Resection and radiotherapy according to the MRI

SUMMARY:
Glioblastoma multiforme (GBM IV WHO) is the most common, primary neoplasm of brain in the adults. Simultanously it is the most agressive one of all primary brain tumors. Despite the treatment the outcome in that group of patients is poor. In case of the optimal therapy the estimated median of survival ranges between 12 and 16 months. The present standard of treatment embraces the gross total resection with the preserved neurological functions and the posoperative management according to the Stupp's protocol (fractionated radiotherapy of 60 Gy dose and the chemotherapy with Temozolamide).

Annually the incidence rate of GBM is 5/100.000 of population. According to the National Tumor Registry 2494 people went down to the malignant neoplasmatic disease of brain classified as C71 (ICD-10) in 2020. The evaluation indicates that it is 600 new patients with the diagnosis of GBM. The disease becomes the 9th cause of death among males and the 13th one among females. The peak of incidence appears in the 5th decade of life and concerns the most productive population. Routinely the management embraces the planning of the resection surgery based on the preoperative magnetic resonance investigation (MRI) with contrast. The common image of the tumor allows to put the preliminary diagnosis with the high probability rate. The GBM occurs as the enhanced tumor with the central necrosis and the circumferential brain edema visible in T2 and Flair sequences of MRI. Commonly the border of tumor becomes the line of contrast enhancement. The enhances area is the aim of surgical treatment. The lack of the preoperative enhanced area in the postoperative MRI is assumed as the gross total resection (GTR). It has been proved that the range of the resection translates into the overall survival (OS) and the progression free survival (PFS). Despite the resection classified as GTR the relapse in the operated area often occurs. It can be explained by the presence of the glioma stem cells in the surrounding neuronal tissue. They are responsible for the early relapse of GBM. Notably, it is evident that the MRI with contrast becomes the method which does not reveal the proper range of resection with the relevant sensitivity so as to extend PFS and OS. The positron emission tomography (PET) is one of the diagnostic methods having been clinically evaluated. PET assesses the metabolic demand of the neoplasm for the biochemical substrates. That methodology is commonly used in case of severity of the solid tumors. The fluorodeoxyglucose (18-FDG) is the most frequently used. However the high metabolism of glucose within the brain, particularly in the grey matter, 18-FDG has the limitation in the process of planning of the tumor resection. The higher specificity and sensitivity are elicited among the markers including aminoacids, praticularly 11-C methionine (11C-MET). Within the gliomas the higher uptake is observed than in the healthy brain. The range of the contrast enhancement in the MRI covers only 58% of the higher 11C-MET metabolism. Comparing these results with a tumor resection beyond the enhancement area, indicates the necessity of the precise assessment of the proposed method in the routine planning of the glioma resection.

Current body of literature lacks in high quality research concerning that issue. The articles regarding the glioma resection beyond the GTR may be found instead. The surgery is limited to the resection of brain area with the incorrect signal in the FLAIR sequence, suspected of the presence of glioma stem cells. The described technique allows to extend PFS by for about 2 months. In that case the resection is based mainly on the FLAIR sequence which does not determine the presence of the neoplasm therein. The fusion of the MRI and the MET-PET images would allow to plan the resection so as to cover the area of incorrectly increased marker uptake.

ELIGIBILITY:
Inclusion Criteria:

* Single macroscopic tumor focus with the appearance of glioblastoma multiforme on MRI with contrast - contrast-enhancing lesion, completely or with central necrosis, with surrounding edema.
* No history of cancer in other organs. No suspicious lesions on X-ray of the chest and abdomen (CT with contrast).
* No clinical suspicion of brain abscess - no meningeal symptoms, signs of neuroinfection, fever, elevated inflammatory parameters.
* Primary tumor, without neurosurgical, radiotherapy or oncology intervention. Prior tumor biopsy is allowed.
* Tumor eligible for surgical treatment - craniotomy and tumor resection.
* Age ≥ 18 years but < 70 years old.
* Quality of life assessment: KPS ≥ 70.
* Informed patient consent to the study and proposed treatment.
* No allergy to contrast agents used in PET and MRI.
* No medical contraindications to neurosurgery - craniotomy and resection.

Exclusion Criteria:

* Multifocal brain tumor.
* Recurrence of glioblastoma multiforme.
* Clinical or radiological suspicion of brain metastasis or brain abscess.
* Postoperative histopathological diagnosis other than WHO grade IV glioblastoma.
* Medical contraindications to any surgery under general anesthesia.
* Pregnancy, breastfeeding.
* Known allergy to gadolinium contrast or radiopharmaceutical tracing agent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2029-07-31 (Estimated); Study Completion 2032-07-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 36 months post surgery
Overall survival | 36 months post surgery

SECONDARY OUTCOMES:
Assessment of tumor volume (GTV) in MRI with contrast in relation to the tumor borders in PET-CT | 1 day before radiotherapy
  It will be assessed as the ratio of the treated tumor volume volumetrically based on MRI+T1C and FLAIR examination by software to the tumor volume estimated in a homogeneous way based on PET-CT examination. Both measurements will be verified independently by a neurosurgeon and a nuclear medicine specialist. This value will allow you to estimate how large the differences are treatment planning based on two different modalities - morphological assessment of the tumor and assessment of metabolic activity.
Volumetric assessment of the planned radiotherapy volume based on PET-MRI and MRI planning. | 1 day before radiotherapy
Long-term survival rate and prognostic factors (longer than 1 year from diagnosis). | 36 months post surgery
  Detailed analysis of factors prognostically favorable for long-term survival, which will allow for better selection of therapeutic options and possible reoperation in this group of patients.
Pattern of local recurrence based on postoperative PET-MRI. Assessment of the nature and location of local recurrence based on the postoperative SUV parameter MET-PET and MRI examination. | 36 months post surgery
  The purpose of this analysis is to develop risk factors for recurrence based on postoperative radiological examinations.
Assessment of quality of life related (SF-36 questionnaire) to the increase in the volume of the tumor undergoing treatment. | 7 days post surgery, 1 day before and after radiotherapy
  Increasing the scope surgery and radiotherapy treatment may result in deterioration of the patient's functioning. Therefore, the above factors will be analyzed for correlation the scope of resection and the functioning of patients. The evaluation will be performed by neurosurgeons and a psychologist trained in neuropsychological assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Kamil Krystkiewicz, PhD, Principal Investigator — Department of Neurosurgery and Neurooncology, Copernicus Memorial Hospital in Łódź, Poland
Locations (1):
- Copernicus Memorial Hospital in Łódź, Poland, Lodz, Łódź Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Herholz K, Holzer T, Bauer B, Schroder R, Voges J, Ernestus RI, Mendoza G, Weber-Luxenburger G, Lottgen J, Thiel A, Wienhard K, Heiss WD. 11C-methionine PET for differential diagnosis of low-grade gliomas. Neurology. 1998 May;50(5):1316-22. doi: 10.1212/wnl.50.5.1316. PMID 9595980
- [Background] Kracht LW, Miletic H, Busch S, Jacobs AH, Voges J, Hoevels M, Klein JC, Herholz K, Heiss WD. Delineation of brain tumor extent with [11C]L-methionine positron emission tomography: local comparison with stereotactic histopathology. Clin Cancer Res. 2004 Nov 1;10(21):7163-70. doi: 10.1158/1078-0432.CCR-04-0262. PMID 15534088
- [Background] Singhal T, Narayanan TK, Jain V, Mukherjee J, Mantil J. 11C-L-methionine positron emission tomography in the clinical management of cerebral gliomas. Mol Imaging Biol. 2008 Jan-Feb;10(1):1-18. doi: 10.1007/s11307-007-0115-2. Epub 2007 Oct 24. PMID 17957408
- [Background] Grosu AL, Weber WA, Riedel E, Jeremic B, Nieder C, Franz M, Gumprecht H, Jaeger R, Schwaiger M, Molls M. L-(methyl-11C) methionine positron emission tomography for target delineation in resected high-grade gliomas before radiotherapy. Int J Radiat Oncol Biol Phys. 2005 Sep 1;63(1):64-74. doi: 10.1016/j.ijrobp.2005.01.045. PMID 16111573
- [Background] Galldiks N, Niyazi M, Grosu AL, Kocher M, Langen KJ, Law I, Minniti G, Kim MM, Tsien C, Dhermain F, Soffietti R, Mehta MP, Weller M, Tonn JC. Contribution of PET imaging to radiotherapy planning and monitoring in glioma patients - a report of the PET/RANO group. Neuro Oncol. 2021 Jun 1;23(6):881-893. doi: 10.1093/neuonc/noab013. PMID 33538838
- [Background] Pirotte B, Goldman S, Dewitte O, Massager N, Wikler D, Lefranc F, Ben Taib NO, Rorive S, David P, Brotchi J, Levivier M. Integrated positron emission tomography and magnetic resonance imaging-guided resection of brain tumors: a report of 103 consecutive procedures. J Neurosurg. 2006 Feb;104(2):238-53. doi: 10.3171/jns.2006.104.2.238. PMID 16509498

DOCUMENTS (1):
  • Informed Consent Form (2022-05-16): https://cdn.clinicaltrials.gov/large-docs/31/NCT06466031/ICF_000.pdf